CLINICAL TRIAL: NCT00467155
Title: Genotypes of Helicobacter Pylori in West African Children and Adults: Part 2: The Application of a Minimally Invasive Technique for H. Pylori Isolation in a Population Study
Brief Title: Helicobacter in The Gambia (Part 2)
Status: Withdrawn | Type: Observational
Sponsor: Medical Research Council Unit, The Gambia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Professor Richard Adegbola, Principal Inestigator, Medical Research Council, Gambia
Other Study IDs: 06-0004
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-04

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori, children, infants, Gambia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine Helicobacter pylori bacteria in the stomach fluids of children who are hospitalized and receiving nutritional care via nasogastric feeding (tube from the nose to the stomach) to treat malnutrition. The H. pylori strains from Gambian children may differ genetically from the strains found in the stomachs of adults from the same community. The fluid samples will be examined for H. pylori bacterial infections that may make children sick and unable to absorb food. Ninety hospitalized Gambian children, less than 2 years of age, requiring a nasogastric feeding tube will have stomach fluid samples taken via the gastric tube. Thirty mothers of children who are positive for H. pylori bacteria will provide a sample of stomach fluid. This study may help develop treatments to heal the stomach and improve child growth. This study will be conducted at the Medical Research Council of Great Britain Research Laboratories and Clinical Facility in Fajara.

DETAILED DESCRIPTION:
This preliminary descriptive study is aimed at providing the first data that will evaluate differences and similarities in genotype between isolates of H. pylori obtained from children and adults living in The Gambia, West Africa, and to assess the likely magnitude of these differences. This protocol describes the application of minimally invasive techniques for H. pylori isolation (developed in the first part of this project and described in a separate protocol, DMID protocol 06-0053) in a population study. Study subjects will be residents of The Gambia, West Africa. Ninety children, aged less than 2 years, requiring therapeutic nasogastric intubation and 30 healthy mothers of these children will be studied. Subjects will be studied at the Medical Research Council (MRC) of Great Britain Research Laboratories and Clinical Facility in Fajara, The Gambia, West Africa. Investigators propose that the transition from childhood colonization to adult disease state is affected by multiple factors including evolution of genotypes of colonizing H. pylori strains themselves, driven in part by the host response to infection. Researchers hypothesize that H. pylori strains from Gambian children will differ genetically from the strains of chronically colonized adults from the same community. The investigators' genetic and phenotypic characterization of pediatric and adult isolates will test for fundamental differences between strains circulating in these 2 age groups, which may help to evaluate the importance of strain selection and/or genome evolution in such high risk societies. The specific aim of this study is to assess the relatedness of child strains and those from close adult relatives. Study procedures will include aspirating gastric juice through a nasogastric tube used for infant feeding purposes in children who are undergoing intensive in-patient re-nutrition, and culturing H. pylori from these aspirates, and also from parents who accept the invitation to donate a sample of gastric juice for culture through a nasogastric tube inserted temporarily for this purpose. Most genotyping will entail arbitrarily primed polymerase chain reaction DNA fingerprinting, limited (focused) DNA sequencing, especially in cases of isolates with closely related but non-identical fingerprints, and metronidazole susceptibility tests. Genetic and phenotypic characterization of pediatric and adult isolates will test for fundamental differences between strains circulating in these two age groups, and thereby help evaluate the importance of strain selection and/or genome evolution in such high risk societies. Subjects will be studied only once during this 2-year project. If H. pylori are isolated from gastric aspirates, the mother of that child will be asked if they would agree to have a nasogastric tube passed on one occasion to obtain an aspirate of gastric juice for H. pylori culture. The isolates obtained will be subject to DNA analysis and genotyping. Specific points to be addressed by these comparative studies will include direct comparison of strains isolated from children and adults from within the same family or village. This will be the first study to be performed in a society with a high early incidence of naturally acquired H. pylori colonization, and will allow direct comparison between isolates from children and adults from within the same families or village environment, which will provide information about intra-familial and intra-community transmission of infection. The main outcome measure is the degree of relatedness between the bacterial isolates. This will be assessed by visual comparison between random amplification of polymorphic DNA (RAPD) results, by comparison of genotype for alleles of interest, and definitively by sequencing of housekeeping genes to construct phylogenetic trees of relatedness using the STAR program and multiple locus sequence typing (MLST) database. There are no outcome measures for human subjects.

ELIGIBILITY:
Inclusion Criteria:

Children: All children under the age of 2 years who are inpatients on the MRC ward and who have a nasogastric tube in situ for the purposes of re-nutrition or other medical management, will be eligible for inclusion. Children must be positive for H. pylori. No lower age limit is specified for the purposes of this study, but an audit of clinical cases shows that all children admitted to the MRC ward who would be eligible for inclusion are aged over 3 months. Children aged under 3 months will not be enrolled.

Adults: Mothers of H. pylori positive children will be eligible for inclusion. In The Gambia subjects aged 18 years and above are considered as adult.

Subjects will be sampled only once.

Subjects cannot be included if they do not agree to provide Informed Consent

Exclusion Criteria:

The use of antibiotics during the 2 weeks prior to recruitment will exclude subjects from the study. Subjects who have participated in any other clinical trial within the last 30 days will be excluded

Ages: 3 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of rural subsistence farmers and semi-urban dwellers attending the clinic at the MRC research laboratories in Fajara, The Gambia. Subjects will comprise; i) children who have a nasogastric tube inserted for nutritional rehabilitation on the ward at Fajara; ii) mothers of children who are found to be H. pylori positive.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
The degree of relatedness between bacterial isolates
  This will be assessed by visual comparison between RAPD results, by comparison of genotypes for alleles of interest, and definitively by sequencing of housekeeping genes to construct phylogenetic trees of relatedness, using the STAR program (a computer program for putting DNA sequences together for analysis) and MLST database.